CLINICAL TRIAL: NCT07385430
Title: Phase 1 Study of LGW16-03 To Identify Nerves
Brief Title: Study of LGW16-03 To Identify Nerves
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eric R. Henderson (Other)
Collaborators: Oregon Health and Science University (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Eric R. Henderson, Assistant Professor, Dartmouth-Hitchcock Medical Center
Organization: Dartmouth-Hitchcock Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 02003082
Record Dates: First submitted 2026-01-13; First posted 2026-02-04 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Adults; Open-field Surgery; Major Nerve
Keywords: Surgery; Nerve; Fluorescence imaging

STUDY DESIGN:
Intervention Model Description: This study is a single-arm, open-label study of LGW16-03.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LGW16-03 (Experimental): Participants will receive a single IV infusion of the investigational drug (LGW16-03).
  Interventions: Drug: LGW16-03

INTERVENTIONS:
Drug: LGW16-03 — LGW16-03 is a non-biological medical imaging agent classified as a contrast agent, consistent with FDA definitions. It is intended to improve intraoperative visualization of specific tissues-namely, peripheral nerves-by enhancing the relative difference in fluorescence signal intensity between nerve and adjacent tissues.

SUMMARY:
The primary goal of this study is to determine the safety and tolerability of LGW16-03, a novel nerve-labeling fluorophore, in participants undergoing open-field orthopaedic surgery. Secondary goals include: 1) identifying the lowest dose without adverse events that provides peak florescence imaging contrast, and 2) characterizing the pharmacokinetics of LGW16-03.

Participants will receive a one-time intravenous infusion of the investigational drug (LGW16-03) prior to their planned surgery. Participants' vitals will be closely monitored and will have blood samples taken at regular intervals. Fluorescence images of their major nerve will be taken during surgery. Participants will have one study follow-up visit approximately 30 days after their surgery.

DETAILED DESCRIPTION:
This is a single-arm, open-label phase I study of LGW16-03, a novel nerve-labeling fluorophore created with the goal of reducing iatrogenic injury to nerves during medical procedures. This study will be conducted in two parts. Part 1-dose escalation- will follow a 3+3 dose-escalation trial design and we will investigate the safety of LGW16-03; pharmacokinetic and fluorescence contrast data will also be collected. Escalation will be stopped if dose-limiting toxicity (DLT) is encountered. Part 2-dose expansion-will continue safety and pharmacokinetic data collection and evaluate further the fluorescence contrast to inform dose. Eligible participants will be limited to healthy patients scheduled for open-field orthopaedic surgical procedures involving exposure of a major compound nerve (i.e., a named nerve with both motor and sensory function). Participants who are determined eligible and who provide informed consent will be administered a single intravenous dose of LGW16-03 on the day of surgery (D0) approximately 60-120 minutes before anticipated induction of anesthesia. Surgical procedures will be conducted per standard of care (SOC) and LGW16-03 will not be used for surgical decision-making. Intraoperative fluorescence imaging (iFI) will begin at the time of first exposure of the target nerve and will be repeated at approximately 30 +/- 15-minute intervals until the target nerve is no longer visible, or the procedure concludes. Imaging will be performed using an FDA-approved fluorescence imaging system (Zeiss Kinevo). At each time point, images of the exposed nerve and adjacent tissues-including muscle, adipose (fat), vasculature, fascia, skin, and/or tendon-will be captured and analyzed for fluorescence signal intensity. These data will be used to calculate nerve-to-background tissue ratios (NBTR) at each time point during the surgery. These data will provide assessment of LGW16-03's ability to provide clinically meaningful intraoperative illumination of the nerve relative to surrounding tissues at the doses being investigated. Additional data will be collected in the form of surveys completed: 1) in real time by the operating surgeon performing trial operations; and 2) surgeons shown images obtained during the surgery who are then asked about the conspicuity of nerve tissue. Up to 24 patients will take part in Part 1, up to 14 patients will take part in Part 2; a maximum of 38 patients will be enrolled in the entire study. Enrollment is expected to take <18 months. Total time for this protocol is estimated to be 24 months.

ELIGIBILITY:
Inclusion Criteria (All of the following criteria must be met by study participants to be eligible for study enrollment):

1. Scheduled and medically cleared for a standard of care, open-field (not endoscopic) surgical procedure wherein a major nerve will be exposed and visible to the imaging equipment.
2. Participants must be willing and able to provide informed consent for participation in the study and adhere to all study procedures.
3. Intact motor and sensory function in the nerve to be imaged, as determined by physical exam performed by the operating surgeon or clinician on the study team, including:

   1. 5/5 motor strength in relevant muscle groups.
   2. Normal sensation on testing with a 5.07 Semmes-Weinstein filament or other valid testing method.
   3. No documented history of neuropathy of any kind.
4. Age ≥ 18 years old.
5. Medical clearance for surgery provided by a supervising medical provider (surgeon or primary care provider).
6. Adequate renal function defined as creatinine clearance ≥ 60mL/min.
7. Adequate liver function:

   1. Total bilirubin ≤ 1.5 x ULN (≤ 3.0 x ULN in patients with Gilbert's disease)
   2. ALT and AST ≤ 2.5 x ULN if no active liver involvement or ALT and AST ≤ 5 xULN with active liver involvement
   3. Albumin ≥3 g/dL
8. Adequate hematologic and clotting function:

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   2. Platelet count ≥ 100 x 109/L
   3. Hemoglobin ≥ 8 g/dL or ≥ 5.6 mmol/L
   4. International Normalized Ratio (INR) ≤ 1.5 x ULN
9. No growth factor support, transfusions, or albumin administration within 14 days of first dose of study treatment
10. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures
11. If of childbearing potential, must have a negative urine or serum pregnancy test and be using a medically acceptable form of contraception (e.g., hormonal birth control, intrauterine devices, double-barrier method) or abstinence.

Exclusion Criteria (Any of the following criteria would exclude a participant from study enrollment):

1. Pregnant or breastfeeding persons who are not willing to stop breastfeeding. Due to the unknown safety profile of LGW16-03 in humans, and the potential for fetal or neonatal exposure through transplacental transfer or breast milk, breastfeeding is not allowed throughout the study and until at least 60 days after last dose.
2. Nerve injury or dysfunction of any kind in the nerve to be imaged (e.g., diabetic neuropathy, multiple sclerosis, other neuropathy, traumatic nerve injury)
3. Peripheral vascular disease requiring management a vascular surgeon.
4. Prior surgery in the planned surgical region within the previous 365 days.
5. Abnormal cardiac rhythm not controlled with medication, history of stroke, coronary events and/or heart failure within 1 year.
6. Current evidence of renal or liver disease.
7. History of fluorescein allergy.
8. Direct administration of a local anesthetic agent in the region of the nerve to be imaged that could affect the motor or sensory function of the target nerve.
9. Any other criteria deemed by the Principal Investigator that may prevent the participant from successfully completing the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Assess safety and tolerability of LGW16-03 | Immediately after infusion of the drug until the post-operative follow-up appointment which will occur approximately 30 days after surgery.
  This study's primary outcome is safety, which will be evaluated by the occurrence of treatment-related adverse events, with attention to frequency and severity as determined by CTCAE v5.0.

SECONDARY OUTCOMES:
Assess dose of LGW16-03 | Immediately after infusion of the drug until the post-operative follow-up appointment which will occur approximately 30 days after surgery.
  This study's first secondary outcome is study drug dose, which will be evaluated by identifying the lowest dose that provides useful fluorescence contrast, which is measured via the nerve-to-background fluorescence contrast ratio.
Assess time of peak LGW16-03 concentration | Regular blood draws will occur from infusion to 24 hours post-infusion.
  The study's second secondary outcome is to assess time of peak LGW16-03 concentration in plasma (Cmax) following intravenous LGW16-03 infusion (hours).

OTHER OUTCOMES:
Evaluate the ability of LGW16-03 to generate detectable fluorescence signal in exposed nerve tissue during surgery. | From when major nerve is first visible during surgery, approximately every 30 minutes until surgery ends.
  Using the Kinevo 900 imager (Carl Zeiss AG, Germany; FDA-approved fluorescence imaging system), fluorescence images will be taken of the surgical field at regular intervals.
Assess operating surgeon-reported experience in identifying nerve tissue with LGW16-03 | Operating surgeon experience will be evaluated immediately following surgery.
  Visual-analog scale (VAS)-based questions of nerve visualization
Assess operating surgeon-reported experience in identifying nerve tissue with LGW16-03 | Operating surgeon experience will be evaluated immediately following surgery.
  Likert scale-based questions of nerve visualization
Assess operating surgeon-reported experience in identifying nerve tissue with LGW16-03 | Operating surgeon experience will be evaluated immediately following surgery.
  Task load index (NASA-TLX) scores, where higher scores indicate higher task load.
Assess non-operating surgeon feedback on identifying nerve tissue with LGW16-03 | Non-operating surgeon feedback will be collected at regular intervals from enrollment through 18 months.
  Visual-analog scale (VAS)-based questions of nerve visualization
Assess non-operating surgeon feedback on identifying nerve tissue with LGW16-03 | Non-operating surgeon feedback will be collected at regular intervals from enrollment through 18 months.
  Likert scale-based questions of nerve visualization
Assess non-operating surgeon feedback on identifying nerve tissue with LGW16-03 | Non-operating surgeon feedback will be collected at regular intervals from enrollment through 18 months.
  Task load index (NASA-TLX) scores, where higher scores indicate higher task load.

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koller M, Qiu SQ, Linssen MD, Jansen L, Kelder W, de Vries J, Kruithof I, Zhang GJ, Robinson DJ, Nagengast WB, Jorritsma-Smit A, van der Vegt B, van Dam GM. Implementation and benchmarking of a novel analytical framework to clinically evaluate tumor-specific fluorescent tracers. Nat Commun. 2018 Sep 18;9(1):3739. doi: 10.1038/s41467-018-05727-y. PMID 30228269
- [Background] National Cancer Institute., Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0, D.o.H.a.H. Services, Editor. 2017, National Institutes of Health, National Cancer Institute: Bethesda, MD.
- [Background] Hart, S.G. and L.E. Staveland, Development of NASA-TLX (Task Load Index): Results of empirical and theoretical research. Advances in Psychology, 1988. 52: p. 139-183.
- [Background] Lowndes BR, Forsyth KL, Blocker RC, Dean PG, Truty MJ, Heller SF, Blackmon S, Hallbeck MS, Nelson H. NASA-TLX Assessment of Surgeon Workload Variation Across Specialties. Ann Surg. 2020 Apr;271(4):686-692. doi: 10.1097/SLA.0000000000003058. PMID 30247331
- [Background] Henderson ER, Elliott J, Jiang S, Gitajn IL, Lee J, Gibbs S, Bouvet M, Mahadevan-Jansen A, Daly M, Streeter SS, Paulsen KD, Pogue BW, Samkoe KS, Singhal S. Proceduralist criteria for evaluating interface utility of novel imaging modalities in early phase clinical trials: evaluating the need for standardized criteria. Proc SPIE Int Soc Opt Eng. 2023 Jan-Feb;12361:123610F. doi: 10.1117/12.2650756. Epub 2023 Mar 14. PMID 37034554
- [Background] Ahlering TE, Eichel L, Skarecky D. Evaluation of long-term thermal injury using cautery during nerve sparing robotic prostatectomy. Urology. 2008 Dec;72(6):1371-4. doi: 10.1016/j.urology.2007.11.101. Epub 2008 Mar 3. PMID 18313123
- [Background] Echeverri A, Flexon PB. Electrophysiologic nerve stimulation for identifying the recurrent laryngeal nerve in thyroid surgery: review of 70 consecutive thyroid surgeries. Am Surg. 1998 Apr;64(4):328-33. PMID 9544143
- [Background] Li R, Liu Z, Pan Y, Chen L, Zhang Z, Lu L. Peripheral nerve injuries treatment: a systematic review. Cell Biochem Biophys. 2014 Apr;68(3):449-54. doi: 10.1007/s12013-013-9742-1. PMID 24037713
- [Background] Zhang J, Moore AE, Stringer MD. Iatrogenic upper limb nerve injuries: a systematic review. ANZ J Surg. 2011 Apr;81(4):227-36. doi: 10.1111/j.1445-2197.2010.05597.x. Epub 2010 Dec 23. PMID 21418465
- [Background] Burke S, Shorten GD. When pain after surgery doesn't go away.. Biochem Soc Trans. 2009 Feb;37(Pt 1):318-22. doi: 10.1042/BST0370318. PMID 19143655
- [Background] Gangadharan S, Sarkaria IN, Rice D, Murthy S, Braun J, Kucharczuk J, Predina J, Singhal S. Multiinstitutional Phase 2 Clinical Trial of Intraoperative Molecular Imaging of Lung Cancer. Ann Thorac Surg. 2021 Oct;112(4):1150-1159. doi: 10.1016/j.athoracsur.2020.09.037. Epub 2020 Nov 19. PMID 33221195
- [Background] Randall LM, Wenham RM, Low PS, Dowdy SC, Tanyi JL. A phase II, multicenter, open-label trial of OTL38 injection for the intra-operative imaging of folate receptor-alpha positive ovarian cancer. Gynecol Oncol. 2019 Oct;155(1):63-68. doi: 10.1016/j.ygyno.2019.07.010. Epub 2019 Jul 27. PMID 31362825
- [Background] Predina JD, Newton AD, Keating J, Dunbar A, Connolly C, Baldassari M, Mizelle J, Xia L, Deshpande C, Kucharczuk J, Low PS, Singhal S. A Phase I Clinical Trial of Targeted Intraoperative Molecular Imaging for Pulmonary Adenocarcinomas. Ann Thorac Surg. 2018 Mar;105(3):901-908. doi: 10.1016/j.athoracsur.2017.08.062. Epub 2018 Feb 15. PMID 29397932
- [Background] Hoogstins CE, Tummers QR, Gaarenstroom KN, de Kroon CD, Trimbos JB, Bosse T, Smit VT, Vuyk J, van de Velde CJ, Cohen AF, Low PS, Burggraaf J, Vahrmeijer AL. A Novel Tumor-Specific Agent for Intraoperative Near-Infrared Fluorescence Imaging: A Translational Study in Healthy Volunteers and Patients with Ovarian Cancer. Clin Cancer Res. 2016 Jun 15;22(12):2929-38. doi: 10.1158/1078-0432.CCR-15-2640. PMID 27306792
- [Background] Stummer W, Pichlmeier U, Meinel T, Wiestler OD, Zanella F, Reulen HJ; ALA-Glioma Study Group. Fluorescence-guided surgery with 5-aminolevulinic acid for resection of malignant glioma: a randomised controlled multicentre phase III trial. Lancet Oncol. 2006 May;7(5):392-401. doi: 10.1016/S1470-2045(06)70665-9. PMID 16648043
- [Background] Orcutt KD, Slusarczyk AL, Cieslewicz M, Ruiz-Yi B, Bhushan KR, Frangioni JV, Wittrup KD. Engineering an antibody with picomolar affinity to DOTA chelates of multiple radionuclides for pretargeted radioimmunotherapy and imaging. Nucl Med Biol. 2011 Feb;38(2):223-33. doi: 10.1016/j.nucmedbio.2010.08.013. Epub 2010 Oct 27. PMID 21315278
- [Background] Vahrmeijer AL, Hutteman M, van der Vorst JR, van de Velde CJ, Frangioni JV. Image-guided cancer surgery using near-infrared fluorescence. Nat Rev Clin Oncol. 2013 Sep;10(9):507-18. doi: 10.1038/nrclinonc.2013.123. Epub 2013 Jul 23. PMID 23881033
- [Background] Gibbs-Strauss SL, Vooght C, Fish KM, Nasr KA, Siclovan TM, Barnhardt NE, Tan Hehir CA, Frangioni JV. Molecular imaging agents specific for the annulus fibrosus of the intervertebral disk. Mol Imaging. 2010 Jun;9(3):128-40. PMID 20487679
- [Background] Frangioni JV. In vivo near-infrared fluorescence imaging. Curr Opin Chem Biol. 2003 Oct;7(5):626-34. doi: 10.1016/j.cbpa.2003.08.007. PMID 14580568